CLINICAL TRIAL: NCT01152229
Title: Platelet Reactivity In Patients With Nuisance Bleeding On A Thienopyridine
Acronym: PLACID
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Michael Gaglia, MD, Cardiovascular Research Institute/ Medstar Health Research Institute
Other Study IDs: PLACID
Record Dates: First submitted 2010-05-28; First posted 2010-06-29 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Platelet Aggregation; Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- nuisance bleeding
- alarming bleeding
- maintenance therapy

SUMMARY:
The objective is to describe and quantify levels of platelet reactivity in three different cohorts of patients taking thienopyridine: patients who report nuisance bleeding, patients who report alarming bleeding, and patients who report no nuisance or alarming bleeding. The investigators hypothesize that patients with nuisance or alarming bleeding events on maintenance thienopyridine therapy will have lower levels of platelet reactivity than patients without nuisance or alarming bleeding on thienopyridine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older from both genders
* Underwent PCI within the last year
* Taking maintenance dose of clopidogrel 75 mg once a day or prasugrel 10 mg once a day for at least five days

Exclusion Criteria:

* Known allergies to aspirin, clopidogrel, or prasugrel.
* Use of a glycoprotein (GP)IIb/IIIa inhibitor within 8 hours of the blood draw.
* Patient known to be pregnant or lactating
* Patient with known history of anemia, thrombocytopenia, bleeding disorder, or currently active bleeding
* On warfarin therapy at the time of blood draw
* Known blood transfusion within the preceding 10 days of the blood draw
* Patients treated with non-steroidal anti-inflammatory drugs (NSAIDS, not to include aspirin) within the previous 5 days
* Any significant medical condition that, in the investigator's opinion, may interfere with the patient's optimal participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone PCI and have reported no bleeding, nuisance bleeding or alarming bleeding.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
platelet reactivity | post percutaneous coronary intervention (PCI) while still on clopidogrel
  Level of platelet reactivity as assessed with the Chrono-Log Lumi-Aggregometer, which measures levels of light transmittance after stimulation with ADP to estimate levels of platelet aggregation.

SECONDARY OUTCOMES:
Platelet reactivity | post PCI while still on clopidogrel
  * Platelet reactivity, as measured with the VerifyNow P2Y12 assay, expressed as platelet reactivity units (PRUs)
  * Platelet reactivity, as assessed with the Vasodilator Stimulated Phosphoprotein (VASP) assay, which measures percentage platelet reactivity inhibition by flow cytometry of the VASP-P protein.
  * Aspirin resistance, as assessed with the VerifyNow aspirin resistance assay, which measures aspirin resistance (ARUs).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gaglia, MD, Principal Investigator — Cardiovascular Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States